CLINICAL TRIAL: NCT01021436
Title: An Open-Label, Multicenter, Multinational Study to Assess the Safety,Tolerability and Pharmacokinetics of Aerosolized Amikacin Delivered Via the Pulmonary Drug Delivery System (NKTR-061) in Intubated and Mechanically- Ventilated Patients With Nosocomial Pneumonia
Brief Title: Safety, Tolerability and Pharmacokinetics of Aerosolized Amikacin in Intubated and Mechanically-ventilated Patients With Nosocomial Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-IN-AK004; 2006-005079-17 (EudraCT Number)
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Pneumonia
Keywords: Pneumonia; Gram-negative bacteria
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amikacin inhalation solution (Experimental): Subjects received 125 mg/mL of aerosolized amikacin via the PDDS clinical device at a nominal dose of 400 mg every 12 h for 7-14 days
  Interventions: Drug: Amikacin inhalation solution (BAY41-6551)

INTERVENTIONS:
Drug: Amikacin inhalation solution (BAY41-6551) — Daily dose of 800 mg of aerosolized amikacin delivered in two divided doses of 400 mg per aerosol treatment 12 hour

SUMMARY:
This study is to understand how the inhaled form of amikacin is spread throughout the human body and how it is eliminated from the body and to make sure that giving an inhaled form of Amikacin to patients is safe and well tolerated

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with confirmed pneumonia, defined as the presence of a new progressive infiltrate(s) on chest radiograph and the presence of gram-negative organism by either culture or Gram stain of respiratory secretions. The subject must be intubated and mechanically ventilated and expected to remain so for at least 3 days after the start of study treatment. Subjects with a tracheostomy were also eligible.

Exclusion Criteria:

* Subjects with compromised or suppressed Immune systems, severe hypoxemia, neutropenia, serum creatinine > 2mg/dl and chronic liver disease
* Had primary lung cancer or another malignancy metastatic to the lungs
* Were known or suspected to have active tuberculosis, cystic fibrosis, acquired immunodeficiency syndrome, or Pneumocystis carinii pneumonia
* Were receiving immunosuppressive therapy, defined as chronic treatment with known immunosuppressant medications
* Had a body mass index of ≥30 kg/m2
* Had burns >40% of total body surface area
* Had known local or systemic hypersensitivity to amikacin or aminoglycosides
* Had a diagnosis of end-stage renal failure or were currently on dialysis treatment
* Had a serum albumin level <2 g/dL at Screening
* Used amikacin by any route within 7 days before the start of study treatment
* Had a presence of any concomitant condition that, in the opinion of the investigator, would preclude completion of study evaluations or make it unlikely that the contemplated course of therapy and Follow-Up could be completed
* Had known respiratory colonization with amikacin-resistant gram-negative rods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Cmax | Pre-dose and up to 12 h post-dose after the start of dosing and also at 1 h and 12 h after the administration of the second dose
  Maximum serum amikacin concentration observed from time 0 to 12 h
Tmax | Pre-dose and up to 12 h post-dose after the start of dosing and also at 1 h and 12 h after the administration of the second dose
  Time that Cmax occurred
AUC0-12h | Pre-dose and up to 12 h post-dose after the start of dosing and also at 1 h and 12 h after the administration of the second dose
  Area under the serum amikacin concentration vs time curve from time 0 to 12 h
Xu0-12h | On Day 3 at the start of dose and up to 12 h after both first and second dose
  Amount of amikacin excreted in urine from 0 to 12 h after dosing
Xu12-24h | On Day 3 at the start of dose and up to 12 h after both first and second dose
  Amount of amikacin excreted in urine from 12 to 24 h after dosing
Xu0-24h | On Day 3 at the start of dose and up to 12 h after both first and second dose
  Amount of amikacin excreted in urine from 0 to 24 h after dosing
Tracheal aspirate | Day 3
Epithelial lining fluid (ELF) concentration | Approximately 15-30 min after completion of the morning dose of study medication on Day 3

SECONDARY OUTCOMES:
Number of participants with adverse events | Approximately 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- United States (4):
  - Birminghan, Alabama
  - Cincinnati, Ohio
  - Memphis, Tennessee
  - Houston, Texas
- France (2):
  - Paris, Cedex 13
  - Limoges, Cedex

REFERENCES:
- [Result] Luyt CE, Clavel M, Guntupalli K, Johannigman J, Kennedy JI, Wood C, Corkery K, Gribben D, Chastre J. Pharmacokinetics and lung delivery of PDDS-aerosolized amikacin (NKTR-061) in intubated and mechanically ventilated patients with nosocomial pneumonia. Crit Care. 2009;13(6):R200. doi: 10.1186/cc8206. Epub 2009 Dec 10. PMID 20003269
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/